CLINICAL TRIAL: NCT01463319
Title: Warm Water Colonoscopy: a Novel Method for Unsedated Colonoscopy
Brief Title: Warm Water and Unsedated Colonoscopy
Acronym: WW
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Presidio Ospedaliero Santa Barbara (Other)
Responsible Party: Principal Investigator, Sergio Cadoni, M.D., Responsabile Servizio Endoscopia Digestiva, Presidio Ospedaliero Santa Barbara
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ASL07_WW-2011
Record Dates: First submitted 2011-10-25; First posted 2011-11-01 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Gastrointestinal Diseases; Digestive System Diseases
Keywords: colonoscopy; warm water method; hydrocolonoscopy; unsedated colonoscopy
MeSH Terms: conditions — Gastrointestinal Diseases; Digestive System Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- warm water irrigation (Experimental): warm water irrigation during insertion phase of colonoscopy
  Interventions: Other: warm water irrigation
- air insufflation (Experimental): air insufflation during insertion phase of colonoscopy
  Interventions: Other: air insufflation

INTERVENTIONS:
Other: air insufflation — air insufflation during insertion phase colonoscopy
  Arms: air insufflation
Other: warm water irrigation — warm water irrigation during insertion phase colonoscopy
  Arms: warm water irrigation

SUMMARY:
Unsedated or slightly sedated colonoscopy has fast recovery time, less cost and lower or no incidence of drug-related side effects. May be slightly painful or discomforting for the patient. Based on numerous recent reports, the investigators designed this randomized controlled trial hypothesizing that the use of warm water irrigation versus air insufflation during the insertion phase of colonoscopy might increase the global tolerability of the examination and the proportion of patients undergoing complete colonoscopy without sedation or with a low dose of sedatives.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 85 Years
* adult patients willing to undergo colonoscopy without routine initial sedation

Exclusion Criteria:

* refuse to initiate colonoscopy without routine sedation
* inadequate bowel preparation
* incapacity to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 818 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
number of patients undergoing complete unsedated or slightly sedated colonoscopy | 9 months
  number of patients undergoing complete unsedated conoloscopy with a pain score (as per used scale) ≤2, or patients with no more than that score AND ≤2 mg Midazolam E.V.

SECONDARY OUTCOMES:
evaluation of pain and tolerability scores | 1 hour
  Numeric rating scale, Verbal Descriptor Scale and Faces Pain Scale (0= no pain, 10 worst possible pain.) Hicks CL et al. Pain 2001;93:173-183. Bieri D. et al. Pain. 1990;41(2):138-50.
percentage of caecum intubation | 1 hour
time to reach caecum | 1 hour
Adenoma detection rate | 9 months
  Proportion of patients with at least one adenoma of any size

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Cadoni, M.D., Principal Investigator — A.S.L. 07 Sardegna
Locations (2):
- Italy (2):
  - Servizio Endoscopia Digestiva, Iglesias, Carbonia-Iglesias
  - U.O.S.D. Diagnostica e Terapia Endoscopica, San Gavino Monreale, Medio Campidano (VS)